CLINICAL TRIAL: NCT00536913
Title: A 4-week, Open-label, Randomized, Multi-centre, Parallel-group Study Evaluating the Safety and Efficacy of 4 Actuations Symbicort® (Budesonide/Formoterol) HFA pMDI 40/2.25 μg Twice Daily, With and Without Spacer, in Children (6-11 Years) With Asthma
Brief Title: Evaluation of Safety and Efficacy of Symbicort® pMDI, With or Without Spacer, in Children (6-11 Years) With Asthma
Acronym: Spacer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5897C00004
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Asthma
Keywords: Symbicort pMDI; spacer; children
MeSH Terms: conditions — Asthma | interventions — Budesonide; Metered Dose Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With Spacer (Experimental): Budesonide/formoterol pMDI 40/2.25ug + spacer
  Interventions: Drug: Budesonide/formoterol pMDI 40/2.25ug + spacer
- Without Spacer (Experimental): Budesonide/formoterol pMDI 40/2.25 ug
  Interventions: Drug: Budesonide/formoterol pMDI 40/2.25 ug

INTERVENTIONS:
Drug: Budesonide/formoterol pMDI 40/2.25ug + spacer
  Arms: With Spacer
Drug: Budesonide/formoterol pMDI 40/2.25 ug
  Arms: Without Spacer

SUMMARY:
The purpose of the study is to compare Symbicort pMDI with and without spacer in terms of steroid potency, improvement of lung function and asthma symptoms in children with asthma (6-11 years).

ELIGIBILITY:
Inclusion Criteria:

* children 6-11 years, diagnosed asthma treated
* 6 months, PEF
* 50% of predicted normal value pre-bronchodilator

Exclusion Criteria:

* current systemic glucocorticosteroids usage
* current respiratory infection
* any significant disease or disorder as judged by investigator

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Anderson, MD PhD, Study Director — AstraZeneca; Piotr Kuna, MD PhD, Principal Investigator — Uniwersytecki Spital
Locations (11):
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kaposvár
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Bytom
  - Research Site, Karpacz
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
- Research Site, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 137 subjects enrolled; 30 non randomised: 26 failed inclusion criteria, 2 voluntary discontinuations, 1 incorrect enrolment, 1 adverse event. 107 subjects were randomised
Period: Overall Study
Arm/Group | With Spacer | Without Spacer
Started | 55 | 52
Completed | 55 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | With Spacer | Without Spacer | Total
Number analyzed (Participants) | 55 | 52 | 107
Age Continuous [Mean (Full Range); unit: years] | 8.6 [6 to 11] | 8.9 [6 to 11] | 8.7 [6 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 34 | 30 | 64

OUTCOME MEASURES:

1. Primary Outcome: Urinary Free Cortisol (UFC)
Description: Ratio between the value at the end of treatment and the value at start of treatment, including only patients with values at both baseline and end of treatment
Time Frame: At baseline and 4 weeks
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | With Spacer | Without Spacer
Number analyzed (Participants) | 54 | 51
Ratio | 0.86 [0.20 to 2.4] | 1.03 [0.12 to 5.4]

2. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Changes in FEV1 from baseline to the mean value at 2 weeks to 4 weeks with the baseline value as a covariate.
Time Frame: At baseline, at 2 weeks and 4 weeks
Measure: Mean (Full Range); unit: Liters
Arm/Group | With Spacer | Without Spacer
Number analyzed (Participants) | 55 | 52
Liters | 0.17 (-0.38) [-0.38 to 0.76] | 0.14 (-0.34) [-0.34 to 0.82]

3. Secondary Outcome: Morning Peak Expiratory Flow (mPEF)
Description: Change in average value from the run-in to the treatment period, calculated using all available data for the 10 last days of run-in, and all available data after randomisation.Missing data between the first and last entry were estimated using linear interpolation.
Time Frame: Daily during run-in and daily during treatment period of 6 weeks
Measure: Mean (Standard Deviation); unit: Liters/min
Arm/Group | With Spacer | Without Spacer
Number analyzed (Participants) | 55 | 52
Liters/min | 28.70 (24.6) | 19.50 (25.1)

4. Secondary Outcome: Evening Peak Expiratory Flow (ePEF)
Description: Change in average value from the run-in to the treatment period, calculated using all available data for the 10 last days of run-in, and all available data after randomisation. Missing data between the first and last entry were estimated using linear interpolation.
Time Frame: Daily during run-in and daily during treatment period of 6 weeks
Measure: Mean (Standard Deviation); unit: Liters/min
Arm/Group | With Spacer | Without Spacer
Number analyzed (Participants) | 55 | 52
Liters/min | 27.00 (27.7) | 15.30 (23.0)

5. Secondary Outcome: Asthma Symptoms at Night
Description: Change in average value from the run-in to treatment period, calculated using all available data for the 10 last days of run-in, and all available data after randomisation.Missing data between the first and last entry estimated using linear interpolation. Daily scale:0 = No symptoms; 1 = Mild symptoms; 2 = Moderate symptoms; 3 = Severe symptoms.
Time Frame: Daily during run-in and daily during treatment period of 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | With Spacer | Without Spacer
Number analyzed (Participants) | 55 | 52
Units on a scale | -0.20 (0.46) | -0.21 (0.39)

6. Secondary Outcome: Asthma Symptoms at Day
Description: as for outcome 5
Time Frame: Daily during run-in and daily during treatment period of 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | With Spacer | Without Spacer
Number analyzed (Participants) | 55 | 52
Units on a scale | -0.25 (0.43) | -0.28 (0.41)

7. Secondary Outcome: Percentage of Nights With Awakenings Due to Asthma
Description: Change in Percentage of nights with awakenings, average value from the run-in to treatment period, calculated using all available data for the 10 last days of run-in, and all available data after randomisation.Missing data between the first and last entry estimated using linear interpolation.
Time Frame: Daily during run-in and daily during treatment period of 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage of nights
Arm/Group | With Spacer | Without Spacer
Number analyzed (Participants) | 55 | 52
Percentage of nights | -13.80 (27.2) | -8.20 (23.8)

8. Secondary Outcome: Use of Rescue Medication at Night
Description: Change in average value from the run-in to treatment period, calculated using all available data for the 10 last days of run-in, and all available data after randomisation.Missing data between the first and last entry estimated using linear interpolation.
Time Frame: Daily during run-in and daily during treatment period of 6 weeks
Measure: Mean (Standard Deviation); unit: Inhalations
Arm/Group | With Spacer | Without Spacer
Number analyzed (Participants) | 55 | 52
Inhalations | -0.21 (0.50) | -0.14 (0.38)

9. Secondary Outcome: Use of Rescue Medication at Day
Description: as for outcome 8
Time Frame: Daily during run-in and daily during treatment period of 6 weeks
Measure: Mean (Standard Deviation); unit: Inhalations
Arm/Group | With Spacer | Without Spacer
Number analyzed (Participants) | 55 | 52
Inhalations | -0.30 (0.56) | -0.19 (0.41)

ADVERSE EVENTS:
Arm/Group | With Spacer | Without Spacer
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/52
Other Adverse Events (participants affected / at risk) | 0/55 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other